CLINICAL TRIAL: NCT01175473
Title: An Open-label, Randomized Two-arm Parallel Group Study to Compare the Effects of 4-week QD Treatment With Lixisenatide or Liraglutide on the Postprandial Plasma Glucose in Patients With Type 2 Diabetes Not Adequately Controlled With Metformin
Brief Title: Effects of Lixisenatide Compared to Liraglutide on the Postprandial Plasma Glucose in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDY10931; 2009-017666-23 (EudraCT Number); U1111-1116-9040 (Other: UTN)
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Liraglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lixisenatide (Experimental): 1-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 2 weeks, followed by 20 mcg QD for up to Week 4.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Metformin
- Liraglutide (Active Comparator): 2-step initiation regimen of liraglutide: 0.6 milligram (mg) QD subcutaneously for 1 week, followed by 1.2 mg QD for 1 week, then 1.8 mg QD up to Week 4.
  Interventions: Drug: Liraglutide; Device: Pre-filled pen injector; Drug: Metformin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self administered by subcutaneous injections once daily 30 minutes before breakfast.
  Arms: Lixisenatide
Device: Pen auto-injector
  Other Names: OptiClik®
  Arms: Lixisenatide
Drug: Liraglutide — Self administered by subcutaneous injections once daily 30 minutes before breakfast.
  Arms: Liraglutide
Device: Pre-filled pen injector
  Other Names: Victoza®
  Arms: Liraglutide
Drug: Metformin — Metformin to be continued at stable dose (1.5 gram per day) up to Week 4.

SUMMARY:
The purpose of the study is to compare the pharmacodynamic effects of lixisenatide (AVE0010), in comparison to liraglutide, as an add-on treatment to metformin, over a period of 4 weeks of treatment.

The primary objective is to assess the effects of lixisenatide, in comparison to liraglutide, in reducing postprandial plasma glucose (PPG) assessed as area under the plasma glucose concentration curve (AUC) after a standardized breakfast at Week 4.

The secondary objectives are to assess the effects of lixisenatide on the maximum PPG excursion, and on the changes in insulin, pro-insulin, C-peptide and glucagon plasma concentrations following a standardized breakfast, 24-hour profile of plasma glucose, glycosylated hemoglobin (HbA1c), satiety markers (obestatin, peptide YY [PYY3-36] and oxyntomodulin); and to assess the clinical and laboratory safety profile.

DETAILED DESCRIPTION:
The duration of the study for each patient is up to 7 weeks including a screening period up to 2 weeks, a treatment period of 4 weeks (Day 1 to Day 28), and an end-of-study visit 7 +/- 2 days after last study drug administration.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes mellitus diagnosed for at least 1 year at the time of screening visit, not adequately controlled by metformin at a dose of at least 1.5 gram per day for at least 3 months prior to screening
* HbA1c greater than or equal to (>=) 6.5% (as recommended by the American Diabetes Association) and HbA1c less than or equal to (<=) 9% at screening
* Covered by Health Insurance System where applicable and/or in compliance with the recommendations of the National (German) Law in force relating to biomedical research
* Not under any administrative or legal supervision

Exclusion criteria:

* At the time of screening age <18 years or >=75 years
* Body Mass Index (BMI): <=20 kilogram per square meter (kg/m^2) or >=37 kg/m^2
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia
* History of myocardial infarction, stroke, or heart failure requiring hospitalization within 6 months prior to the time of screening, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Cardiovascular, hepatic, neurological, or endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult (euthyroid patients on replacement therapy are to be included if the dosage of thyroxin is stable for at least 3 months prior to the screening visit)
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic or diastolic blood pressure >160 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Any clinically significant abnormality identified on physical examination, laboratory tests, or vital signs at the time of screening that in the judgment of the investigator or any sub-investigator precludes safe completion of the study
* Receipt of blood or plasma products within 3 months prior to the time of screening
* Investigator or any sub-investigator, pharmacist, study coordinator, or their study staff or relative thereof directly involved in the conduct of the protocol
* Patients who are considered by the investigator or any sub-investigator as inappropriate for this study for any reason (for example, impossibility of meeting specific protocol requirements such as scheduled visits, being unable to do self-injections, etc.)
* Use of other oral or injectable antidiabetic or hypoglycemic agents other than metformin (for example, alpha glucosidase inhibitor, exenatide, dipeptidyl peptidase IV [DPP-IV] inhibitors, insulin, thiazolidinedione, sulfonylurea, etc.) within 3 months prior to the time of screening
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to the time of screening
* Likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol
* Use of any investigational drug within 3 months prior to screening
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to, gastroparesis and gastroesophageal reflux disease requiring medical treatment within 6 months prior to the time of screening
* Any previous treatment with lixisenatide or liraglutide
* Allergic reaction to any glucagon like peptide - 1 (GLP-1) agonist in the past (for example, exenatide) or to metacresol
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease
* Personal or family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Laboratory findings at the time of screening: alanine aminotransferase: >3 times the upper limit of the normal (ULN) laboratory range; calcitonin >=20 picogram per milliliter (pg/mL); amylase and lipase >3 times ULN; total bilirubin >1.5 times ULN (except in case of Gilbert's syndrome); hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100,000/mm^3; positive test for Hepatitis B surface antigen and/or Hepatitis C antibody and Positive reaction to tests for anti-human immunodeficiency virus (HIV) type 1 (HIV1) and anti-HIV2 antibodies
* Renal impairment defined by creatinine clearance <60 milliliter per minute (mL/min) using the Cockcroft-Gault formula

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Germany (7):
  - Sanofi-Aventis Investigational Site Number 276006, Berlin
  - Sanofi-Aventis Investigational Site Number 276004, Kiel
  - Sanofi-Aventis Investigational Site Number 276002, Mainz
  - Sanofi-Aventis Investigational Site Number 276003, Mannheim
  - Sanofi-Aventis Investigational Site Number 276005, Mönchengladbach
  - Sanofi-Aventis Investigational Site Number 276007, München
  - Sanofi-Aventis Investigational Site Number 276001, Neuss

REFERENCES:
- [Result] Kapitza C, Forst T, Coester HV, Poitiers F, Ruus P, Hincelin-Mery A. Pharmacodynamic characteristics of lixisenatide once daily versus liraglutide once daily in patients with type 2 diabetes insufficiently controlled on metformin. Diabetes Obes Metab. 2013 Jul;15(7):642-9. doi: 10.1111/dom.12076. Epub 2013 Feb 25. PMID 23368510

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 centers in Germany between August 03, 2010 and November 18, 2010.
Pre-assignment Details: A total of 259 patients were screened of which 111 (42.9%) were screen failures. A total of 148 patients were randomized.
Groups:
- Lixisenatide: 1-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) subcutaneously for 2 weeks, followed by 20 mcg QD up to Week 4.
Period: Overall Study
Arm/Group | Lixisenatide | Liraglutide
Started | 77 (Randomized and treated.) | 71
Safety Population | 77 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 71
Pharmacodynamic (PD) Population | 75 (All patients who received at least 1 dose; had baseline and at least 1 post-baseline PD assessment.) | 68
Completed | 75 | 69
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Lixisenatide: 1-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 2 weeks, followed by 20 mcg QD up to Week 4.
- Liraglutide: 2-step initiation regimen of liraglutide: 0.6 mg QD subcutaneously for 1 week, followed by 1.2 mg QD for 1 week, then 1.8 mg QD up to Week 4.
- Total: Total of all reporting groups
Arm/Group | Lixisenatide | Liraglutide | Total
Number analyzed (Participants) | 77 | 71 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (7.5) | 59.7 (8.5) | 60.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 21 | 49
  Male | 49 | 50 | 99
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 76 | 71 | 147
  Black | 1 | 0 | 1
Area Under Plasma Glucose Concentration Curve From Time 0.5 Hours to 4.5 Hours (GLU-AUC0:30-4:30h) [Mean (Standard Deviation); unit: hour*milligram per deciliter (h*mg/dL)] — The area under the plasma glucose concentration time curve (GLU-AUC0:30-4:30h) was calculated using the linear trapezoidal rule from time of breakfast start (8:00 clock time; prior to standardized breakfast [time: 0.5 hours]) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast plasma glucose concentration (time: 0.5 hours). GLU-AUC0:30-4:30h on Day -1 was the baseline. PD population was evaluable for this baseline characteristic.
  hour*milligram per deciliter (h*mg/dL) | 169.41 (84.03) | 183.86 (100.89) | 176.28 (92.39)
Postprandial Plasma Glucose (PPG) Excursion [Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)] — PPG excursion was determined on Day -1 (baseline) as the maximum change in PPG from time of breakfast start (8:00 clock time; prior to standardized breakfast [time: 0.5 hours]) until 4 hours later subtracted from pre-meal plasma concentration. PD population was evaluable for this baseline characteristic.
  milligram per deciliter (mg/dL) | 88.06 (29.31) | 88.06 (35.86) | 88.06 (32.47)
Pro-insulin AUC(0:30-4:30h) [Mean (Standard Deviation); unit: hour*micro international unit/milliliter] — The area under the pro-insulin concentration time curve (AUC0:30-4:30h) was calculated using the linear trapezoidal rule from time of breakfast start (8:00 clock time; prior to standardized breakfast [time: 0.5 hours]) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast pro-insulin concentration (time: 0.5 hours). Pro-insulin AUC0:30-4:30h on Day -1 was the baseline. PD population was evaluable for this baseline characteristic.
  hour*micro international unit/milliliter | 5.68 (6.25) | 6.54 (5.40) | 6.09 (5.86)
Insulin AUC(0:30-4:30h) [Mean (Standard Deviation); unit: hour*micro international unit/milliliter] — The area under the insulin concentration time curve (AUC0:30-4:30h) was calculated using the linear trapezoidal rule from time of breakfast start (8:00 clock time; prior to standardized breakfast [time: 0.5 hours]) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast insulin concentration (time: 0.5 hours). Insulin AUC0:30-4:30h on Day -1 was the baseline. PD population was evaluable for this baseline characteristic.
  hour*micro international unit/milliliter | 99.55 (43.61) | 93.24 (57.30) | 96.55 (50.50)
C-Peptide AUC(0:30-4:30h) [Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)] — The area under the C-peptide concentration time curve (AUC0:30-4:30h) was calculated using the linear trapezoidal rule from time of breakfast start (8:00 clock time; prior to standardized breakfast [time: 0.5 hours]) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast C-peptide concentration (time: 0.5 hours). C-peptide AUC0:30-4:30h on Day -1 was the baseline. PD population was evaluable for this baseline characteristic.
  hour*nanogram per milliliter (h*ng/mL) | 10.61 (4.44) | 9.99 (4.89) | 10.31 (4.65)
Glucagon AUC(0:30-4:30h) [Mean (Standard Deviation); unit: hour*picogram per milliliter (h*pg/mL)] — The area under the glucagon concentration time curve (AUC0:30-4:30h) was calculated using the linear trapezoidal rule from time of breakfast start (8:00 clock time; prior to standardized breakfast [time: 0.5 hours]) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast glucagon concentration (time: 0.5 hours). Glucagon AUC0:30-4:30h on Day -1 was the baseline. PD population was evaluable for this baseline characteristic.
  hour*picogram per milliliter (h*pg/mL) | 27.10 (60.54) | 16.47 (78.98) | 22.05 (69.87)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] — HbA1c on Day 1 (pre-dose [hour 0]) was the baseline. Number of patients analyzed = 74 and 68 for Lixisenatide and Liraglutide arms, respectively.
  percentage of hemoglobin | 7.20 (0.63) | 7.41 (0.81) | 7.30 (0.72)
Peptide YY3-36 (PYY3-36) Concentration [Mean (Standard Deviation); unit: picomole per liter (pmol/L)] — PYY3-36 concentration was determined at 0.5 (8:00 clock time; prior to standardized breakfast), 2.5 and 4.5 hours on Day -1 (time-matched baseline). PD population was evaluable for this baseline characteristic.
  picomole per liter (pmol/L)
    0.5 h | 17.60 (9.46) | 17.83 (9.29) | 17.71 (9.35)
    2.5 h | 21.73 (11.83) | 21.02 (9.19) | 21.40 (10.62)
    4.5 h | 21.98 (10.74) | 20.88 (10.66) | 21.46 (10.68)
Obestatin Concentration [Mean (Standard Deviation); unit: nanomole per liter (nmol/L)] — Obestatin concentration was determined at 0.5 (8:00 clock time; prior to standardized breakfast), 2.5 and 4.5 hours on Day -1 (time-matched baseline). PD population was evaluable for this baseline characteristic.
  nanomole per liter (nmol/L)
    0.5 h | 0.24 (0.12) | 0.29 (0.18) | 0.26 (0.15)
    2.5 h | 0.22 (0.11) | 0.26 (0.15) | 0.24 (0.13)
    4.5 h | 0.24 (0.12) | 0.27 (0.17) | 0.25 (0.15)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Area Under the Plasma Glucose Concentration Curve From Time 0.5 Hours to 4.5 Hours (GLU-AUC0:30-4:30h) at Day 28
Description: The area under the plasma glucose concentration time curve (GLU-AUC0:30-4:30h) was calculated using the linear trapezoidal rule from time of breakfast start (30 minutes after study drug administration [time: 0.5 hours] on Day 28) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast plasma glucose concentration (time: 0.5 hours). GLU-AUC0:30-4:30h on Day -1 was the baseline. Change in GLU-AUC0:30-4:30h = GLU-AUC0:30-4:30h on Day 28 minus GLU-AUC0:30-4:30h on Day -1.
Time Frame: 0.5 (8:00 clock time; prior to standardized breakfast), 0.75, 1, 1.5, 2, 2.5, 3.5, 4.5 hours on Day -1 (baseline), 0.5 (prior to standardized breakfast), 0.75, 1, 1.5, 2, 2.5, 3.5, 4.5 hours post study drug administration on Day 28
Population: Pharmacodynamic (PD) population (modified intent-to-treat [mITT] population) included all randomized patients, who received at least 1 dose of lixisenatide or liraglutide, and had both a baseline assessment and at least 1 post-baseline assessment of any pharmacodynamic variable, irrespective of compliance with the study protocol and procedures.
Measure: Least Squares Mean (95% Confidence Interval); unit: h*mg/dL
Groups:
- Lixisenatide: 1-step initiation regimen of lixisenatide.
- Liraglutide: 2-step initiation regimen of liraglutide.
Arm/Group | Lixisenatide | Liraglutide
Number analyzed (Participants) | 75 | 68
h*mg/dL | -227.25 (120.26) [-246.88 to -207.61] | -72.83 (79.66) [-93.19 to -52.46]
Statistical Analysis 1: Comparison: Lixisenatide vs Liraglutide; To detect a difference of 100 or 150 h*mg/dL in change from baseline to Day 28 in GLU-AUC(0:30-4:30h) between lixisenatide and liraglutide, 60 patients per group would provide a power of 90% assuming common standard deviation of 170 or 250 h*mg/dL, respectively, with a 2-sided test at 5% significance level; Test type: Superiority or Other; p < 0.0001, Linear fixed effects model — Linear fixed effects model with fixed terms for treatment, study site and GLU-AUC(0:30-4:30h) at baseline as covariate was used (using Statistical Analysis System [SAS®] PROC MIXED procedure); No alpha adjustment was performed; Least squares (LS) Mean Difference = -154.42, 95% CI 2-sided [-180.30 to -128.54]

2. Secondary Outcome: Change From Baseline in Postprandial Plasma Glucose (PPG) Excursion at Day 28
Description: PPG excursion was determined on Day -1 (Baseline) and 28 as the maximum change in PPG from time of breakfast start (time: 0.5 hours) until 4 hours later subtracted from pre-meal plasma concentration.
Time Frame: as for outcome 1
Population: PD population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Lixisenatide | Liraglutide
Number analyzed (Participants) | 75 | 68
mg/dL | -70.43 (42.04) [-77.83 to -63.03] | -24.93 (33.67) [-32.57 to -17.29]

3. Secondary Outcome: Change From Baseline in Pro-insulin AUC(0:30-4:30h) at Day 28
Description: The area under the pro-insulin concentration time curve (AUC0:30-4:30h) was calculated using the linear trapezoidal rule from time of breakfast start (30 minutes after study drug administration [time: 0.5 hours] on Day 28) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast pro-insulin concentration (time: 0.5 hours). Pro-insulin AUC0:30-4:30h on Day -1 was the baseline. Change in pro-insulin AUC0:30-4:30h = pro-insulin AUC0:30-4:30h on Day 28 minus pro-insulin AUC0:30-4:30h on Day -1.
Time Frame: 0.5 (8:00 clock time; prior to standardized breakfast), 1, 1.5, 2.5, 3.5, 4.5 hours on Day -1 (baseline), 0.5 (prior to standardized breakfast), 1, 1.5, 2.5, 3.5, 4.5 hours post study drug administration on Day 28
Population: PD population.
Measure: Least Squares Mean (95% Confidence Interval); unit: hour*micro international unit/milliliter
Arm/Group | Lixisenatide | Liraglutide
Number analyzed (Participants) | 75 | 68
hour*micro international unit/milliliter | -1.27 (6.18) [-2.36 to -0.18] | -2.47 (4.86) [-3.59 to -1.34]

4. Secondary Outcome: Change From Baseline in Insulin AUC(0:30-4:30h) at Day 28
Description: The area under the insulin concentration time curve (AUC0:30-4:30h) was calculated using the linear trapezoidal rule from time of breakfast start (30 minutes after study drug administration [time: 0.5 hours] on Day 28) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast insulin concentration (time: 0.5 hours). Insulin AUC0:30-4:30h on Day -1 was the baseline. Change in insulin AUC0:30-4:30h = insulin AUC0:30-4:30h on Day 28 minus insulin AUC0:30-4:30h on Day -1.
Time Frame: as for outcome 3
Population: PD population.
Measure: Least Squares Mean (95% Confidence Interval); unit: hour*micro international unit/milliliter
Arm/Group | Lixisenatide | Liraglutide
Number analyzed (Participants) | 75 | 68
hour*micro international unit/milliliter | -64.22 (59.74) [-78.20 to -50.24] | 5.34 (57.82) [-9.16 to 19.84]

5. Secondary Outcome: Change From Baseline in C-Peptide AUC(0:30-4:30h) at Day 28
Description: The area under the C-peptide concentration time curve (AUC0:30-4:30h) was calculated using the linear trapezoidal rule from time of breakfast start (30 minutes after study drug administration [time: 0.5 hours] on Day 28) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast C-peptide concentration (time: 0.5 hours). C-peptide AUC0:30-4:30h on Day -1 was the baseline. Change in C-peptide AUC0:30-4:30h = C-peptide AUC0:30-4:30h on Day 28 minus C-peptide AUC0:30-4:30h on Day -1.
Time Frame: as for outcome 3
Population: PD population.
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Lixisenatide | Liraglutide
Number analyzed (Participants) | 75 | 68
h*ng/mL | -5.03 (5.97) [-6.33 to -3.72] | 1.04 (4.71) [-0.31 to 2.39]

6. Secondary Outcome: Change From Baseline in Glucagon AUC(0:30-4:30h) at Day 28
Description: The area under the glucagon concentration time curve (AUC0:30-4:30h) was calculated using the linear trapezoidal rule from time of breakfast start (30 minutes after study drug administration [time: 0.5 hours] on Day 28) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast glucagon concentration (time: 0.5 hours). Glucagon AUC0:30-4:30h on Day -1 was the baseline. Change in glucagon AUC0:30-4:30h = glucagon AUC0:30-4:30h on Day 28 minus glucagon AUC0:30-4:30h on Day -1.
Time Frame: as for outcome 3
Population: PD population.
Measure: Least Squares Mean (95% Confidence Interval); unit: h*pg/mL
Arm/Group | Lixisenatide | Liraglutide
Number analyzed (Participants) | 75 | 68
h*pg/mL | -46.71 (67.90) [-61.60 to -31.83] | -25.28 (68.07) [-40.65 to -9.90]

7. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Day 29
Description: Change = HbA1c value at Day 29 (24 hours post-dose on Day 28) minus HbA1c value at baseline (pre-dose [Hour 0] on Day 1).
Time Frame: Pre-dose (Hour 0) on Day 1 and 29 (that is, 24 hours post-dose on Day 28)
Population: PD population. Here, number of patients analyzed = patients with post-baseline HbA1c assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of hemoglobin
Arm/Group | Lixisenatide | Liraglutide
Number analyzed (Participants) | 75 | 67
percentage of hemoglobin | -0.32 (0.30) [-0.40 to -0.24] | -0.45 (0.40) [-0.54 to -0.37]

8. Secondary Outcome: Change From Time-matched Baseline in Peptide YY3-36 (PYY3-36) Concentration at Day 28
Description: Change was calculated by subtracting time-matched baseline value from Day 28 value. Baseline value was the Day -1 time-matched PYY-36 assessment.
Time Frame: 0.5 (8:00 clock time; prior to standardized breakfast), 2.5, 4.5 hours on Day -1 (baseline), 0.5 (prior to standardized breakfast), 2.5, 4.5 hours post study drug administration on Day 28
Population: PD population.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Lixisenatide | Liraglutide
Number analyzed (Participants) | 75 | 68
pmol/L
  Change at Day 28: 0.5 h | 0.02 (5.32) | -0.79 (6.77)
  Change at Day 28: 2.5 h | -7.09 (8.38) | -3.14 (6.67)
  Change at Day 28: 4.5 h | -8.33 (6.73) | -2.47 (7.66)

9. Secondary Outcome: Change From Time-matched Baseline in Obestatin Concentration at Day 28
Description: Change was calculated by subtracting time-matched baseline value from Day 28 value. Baseline value was the Day -1 time-matched obestatin assessment.
Time Frame: as for outcome 8
Population: PD population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Lixisenatide | Liraglutide
Number analyzed (Participants) | 75 | 68
nmol/L
  Change at Day 28: 0.5 h | 0.04 (0.09) | 0.02 (0.11)
  Change at Day 28: 2.5 h | 0.03 (0.09) | 0.01 (0.11)
  Change at Day 28: 4.5 h | -0.01 (0.08) | -0.01 (0.12)

10. Secondary Outcome: Percentages of Patients by Ranges of Oxyntomodulin Levels
Description: Percentage of patients with oxyntomodulin level less than or equal to (<=) limit of detection (LOD), above limit of quantification (LOQ) and between LOD and LOQ were reported. The LOD and LOQ values for oxyntomodulin were 70 and 200 picogram per milliliter (pg/mL) respectively.
Time Frame: as for outcome 8
Population: PD population. Here, 'n' signifies patients with oxyntomodulin assessment at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Liraglutide
Number analyzed (Participants) | 75 | 68
percentage of participants
  Day -1, 0.5 h: <=LOD (n = 75, 68) | 33.3 | 20.6
  Day -1, 0.5 h: LOD-LOQ (n = 75, 68) | 49.3 | 55.9
  Day -1, 0.5 h: >LOQ (n = 75, 68) | 17.3 | 23.5
  Day -1, 2.5 h: <=LOD (n = 75, 68) | 12.0 | 8.8
  Day -1, 2.5 h: LOD-LOQ (n = 75, 68) | 25.3 | 23.5
  Day -1, 2.5 h: >LOQ (n = 75, 68) | 62.7 | 67.6
  Day -1, 4.5 h: <=LOD (n = 75, 68) | 17.3 | 11.8
  Day -1, 4.5 h: LOD-LOQ (n = 75, 68) | 34.7 | 39.7
  Day -1, 4.5 h: >LOQ (n = 75, 68) | 48.0 | 48.5
  Day 28, 0.5 h: <=LOD (n = 75, 68) | 38.7 | 30.9
  Day 28, 0.5 h: LOD-LOQ (n = 75, 68) | 40.0 | 51.5
  Day 28, 0.5 h: >LOQ (n = 75, 68) | 21.3 | 17.6
  Day 28, 2.5 h: <=LOD (n = 74, 68) | 52.7 | 16.2
  Day 28, 2.5 h: LOD-LOQ (n = 74, 68) | 32.4 | 48.5
  Day 28, 2.5 h: >LOQ (n = 74, 68) | 14.9 | 35.3
  Day 28, 4.5 h: <=LOD (n = 75, 68) | 52.0 | 20.6
  Day 28, 4.5 h: LOD-LOQ (n = 75, 68) | 33.3 | 52.9
  Day 28, 4.5 h: >LOQ (n = 75, 68) | 14.7 | 26.5

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration, up to 31 days
Description: Median exposure to study treatment was 28 days in both treatment arms. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Arm/Group | Lixisenatide | Liraglutide
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/71
Other Adverse Events (participants affected / at risk) | 36/77 | 47/71
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (N=77) | Liraglutide (N=71)
Nasopharyngitis (Infections and infestations) | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 14 | 26
Dizziness (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 9 | 11
Abdominal distension (Gastrointestinal disorders) | 5 | 9
Constipation (Gastrointestinal disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 11
Dyspepsia (Gastrointestinal disorders) | 6 | 12
Nausea (Gastrointestinal disorders) | 17 | 16
Vomiting (Gastrointestinal disorders) | 8 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Fatigue (General disorders) | 5 | 4

LIMITATIONS AND CAVEATS:
Data for "Percentages of patients by ranges of oxyntomodulin levels" was reported instead of "Change from Baseline in oxyntomodulin concentration at Day 28" due to change in planned analysis as there were high numbers of values below the LOD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.